CLINICAL TRIAL: NCT03568734
Title: Cesarean Section and Intestinal Flora of the Newborn
Acronym: SECFLOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sture Andersson (Other)
Responsible Party: Sponsor-Investigator, Sture Andersson, Professor, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SECFLOR
Record Dates: First submitted 2017-11-20; First posted 2018-06-26 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Intestinal Microbiome
Keywords: microbiome; transplant; infant; newborn
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: 12 mothers participating in the study (due for caesarean section) are screened for transmissible diseases. A transplant sample is gathered from the mother, processed, and given to the infant at delivery by caesarean section.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transplant arm (Experimental): Fecal transplant sample given to child at delivery
  Interventions: Other: Fecal transplant

INTERVENTIONS:
Other: Fecal transplant — At delivery, i.e. 39-40 weeks of gestation, the newborn infant is given 0.1 g maternal fecal sample (in 0.5 ml of the isotonic saline+10 % glycerol) dissolved in 10 ml of bank milk orally. The sample is given within 2 h of birth. Milk containing fecal sample (2 ml) is given as a part of a total feeding of 5-10 ml.

SUMMARY:
Mode of delivery affects gut microbiome of the infant. Infants born by caesarean section have a less heterogenous microbiome for the first weeks of life. This has been associated with an increased risk for atopy-related diseases, such as allergy and asthma. In this proof-of-principle study the investigators evaluate whether an orally delivered maternal fecal transplant to the infant during the first hours of life affects gut microbiome of the infant

DETAILED DESCRIPTION:
Background

The immune system is affected by the colonizing microbiome. The gut microbiome has been associated with a multitude of inflammatory diseases, such as the development of autoimmune diseases. The association between microbiome and allergic diseases, asthma, type I diabetes and inflammatory bowel diseases have been demonstrated. Moreover, changes in gut microbiome during the first weeks of life have been associated with the development of atopy.

Already at birth, a low concentration of bacteria is present in the meconium of the vaginally delivered infant. Although the neonatal stool is not fully sterile, colonization of the intestinal tract takes place at delivery and throughout the first years of life. The gut microbiome of infants delivered vaginally (VD) and by cesarean section (CS) differs markedly from each other and this difference persists throughout the first years of life. The gut microbiome of infants born by CS have a lower total microbiota diversity and lower Th1 response than those born by VD. Infants delivered by CS been shown to be more likely to develop chronic inflammatory and allergic diseases, eg. inflammatory bowel disease, and systemic connective disorders, and asthma than those delivered vaginally.

Partial restoration of the microbiota of CS-infants was seen when introduced with vaginal microbial transfer. However, the vaginal microbiome is very limited to mainly Lactobacillus spp. and does not contain the microbes that are abundant in the gut microbiota of the mother. Fecal transplantation, or intestinal microbiota transfer, is used to treat chronic infections of Clostridium difficile. However, fecal transplantation has not been used to compensate for the low diversity of CS infants. In this pilot, proof-of-concept and safety evaluation study, the researchers aim to assess the feasibility of fecal transplantation after birth in infants delivered by CS.

ELIGIBILITY:
Inclusion criteria:

* healthy pregnancy
* planned cesarean section delivery

Exclusion criteria:

Maternal exclusion criteria:

* positive GBS status
* maternal refusal
* maternal antibiotic treatment within the last 3 months
* any travel outside of European Union within the last 3 months
* multiple pregnancy and CS after the onset of labor (non-elective CS)

Infant exclusion criteria:

* Apgar score of less than 8
* disturbances of neonatal adaptation (such as transient tachypnea of the newborn)
* antibiotic treatment of the newborn before discharge

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women only
Enrollment: 7 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 0-3 postnatal days
  Clinical condition, inflammatory markers

SECONDARY OUTCOMES:
Attachment of transplant | 1 to 12 weeks of age
  Evaluation of microbiome in comparison to transplant from samples taken from infants weekly at 1-4 weeks of life and at 3 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Sture Andersson, Prof, Principal Investigator — Professor of neonatology
Locations (1):
- Helsinki University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Korpela K, Helve O, Kolho KL, Saisto T, Skogberg K, Dikareva E, Stefanovic V, Salonen A, Andersson S, de Vos WM. Maternal Fecal Microbiota Transplantation in Cesarean-Born Infants Rapidly Restores Normal Gut Microbial Development: A Proof-of-Concept Study. Cell. 2020 Oct 15;183(2):324-334.e5. doi: 10.1016/j.cell.2020.08.047. Epub 2020 Oct 1. PMID 33007265